CLINICAL TRIAL: NCT00907855
Title: Clinical Role of the Duke Activity Status Index in the Selection of the Optimal Type of Stress Myocardial Perfusion Imaging Study in Patients With Known or Suspected Ischemic Heart Disease
Brief Title: Using Duke Activity Status Index (DASI) to Select Optimal Cardiac Stress Tests
Acronym: DASI-08-713
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Lawrence Phillips, MD, Director, Nuclear Cardiology, NYU Langone Health
Other Study IDs: NYU DASI 08-713
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Ischemic Heart Disease
Keywords: Ischemic Heart Disease; Duke Activity Status Index; Stress Myocardial Perfusion Imaging
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cardiac stress testing with functional nuclear imaging is an invaluable technique in the diagnostic and prognostic evaluation of patients with known or suspected ischemic heart disease. Selection of the appropriate type of nuclear stress test: exercise stress Myocardial Perfusion Imaging (MPI) versus pharmacologic stress MPI is crucial for not only diagnostic accuracy and prognostic evaluation, but also for sound clinical decisions and resource utilization.

The Duke Activity Status Index (DASI) is a 12-item questionnaire that utilized self-reported physical work capacity to estimate peak metabolic equivalents (METs) and has been shown to be a valid measurement of functional capacity. The investigators hypothesized that the DASI may be the screening tool that evaluates functional capacity and guides selection of the optimal stress MPI study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred by their primary physician to the Nuclear Lab at NYU School of Medicine for stress myocardial perfusion imaging testing.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-04

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer H. Mieres, MD, Principal Investigator — Division of Cardiology, New York University School of Medicine; Lawrence Phillips, MD, Study Director — Division of Cardiology, New York University School of Medicine
Locations (1):
- Nuclear Cardiology/Stress Lab, NYU Cardiology Division, New York, New York, United States

REFERENCES:
- [Background] Shaw LJ, Olson MB, Kip K, Kelsey SF, Johnson BD, Mark DB, Reis SE, Mankad S, Rogers WJ, Pohost GM, Arant CB, Wessel TR, Chaitman BR, Sopko G, Handberg E, Pepine CJ, Bairey Merz CN. The value of estimated functional capacity in estimating outcome: results from the NHBLI-Sponsored Women's Ischemia Syndrome Evaluation (WISE) Study. J Am Coll Cardiol. 2006 Feb 7;47(3 Suppl):S36-43. doi: 10.1016/j.jacc.2005.03.080. PMID 16458169
- [Background] Hlatky MA, Boineau RE, Higginbotham MB, Lee KL, Mark DB, Califf RM, Cobb FR, Pryor DB. A brief self-administered questionnaire to determine functional capacity (the Duke Activity Status Index). Am J Cardiol. 1989 Sep 15;64(10):651-4. doi: 10.1016/0002-9149(89)90496-7. PMID 2782256